CLINICAL TRIAL: NCT00611533
Title: A Controlled Trial of Atomoxetine in the Treatment of Mild to Moderate Cognitive Difficulties in Menopausal Women
Brief Title: Placebo Controlled Study of Atomoxetine in the Treatment of Mild to Moderate Cognitive Difficulties in Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0403026533
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Menopause; Cognitive Disturbances
Keywords: Menopause; Cognition
MeSH Terms: conditions — Cognition Disorders | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atomoxetine (Active Comparator): Subjects were enrolled into a double-blind, placebo-controlled cross over study where they will receive ATX 40mg/d x 1 week, then 80mg/d x 5 weeks or placebo (PBO) for 6 weeks, followed by a 4-week wash out period that is followed by an additional 6 weeks of treatment in the alternate condition. The 4-week washout period include a 4-day taper in the first week. Subjects undergo assessments of cognition, mood, and menopausal symptoms prior to randomization, after 6 weeks in the first treatment condition (ATX or PBO) and then finally after the second 6-week period of the alternate treatment condition. Subjects are monitored every other week to assess medication compliance and side effects. Subjects will be instructed to take one capsule of ATX 40mg/d or placebo per day. If tolerated, the number of pills of ATX will be increased to 2 per day at the end of Week 1 of both Trials A and B. Subjects will remain on two capsules per day for the remaining 5 weeks of Trials A and B.
  Interventions: Drug: atomoxetine
- Placebo (Placebo Comparator): Subjects were enrolled into a double-blind, placebo-controlled cross over study where they will receive ATX 40mg/d x 1 week, then 80mg/d x 5 weeks or placebo (PBO) for 6 weeks, followed by a 4-week wash out period that is followed by an additional 6 weeks of treatment in the alternate condition. The 4-week washout period include a 4-day taper in the first week. Subjects undergo assessments of cognition, mood, and menopausal symptoms prior to randomization, after 6 weeks in the first treatment condition (ATX or PBO) and then finally after the second 6-week period of the alternate treatment condition. Subjects are monitored every other week to assess medication compliance and side effects. Subjects will be instructed to take one capsule of ATX 40mg/d or placebo per day. If tolerated, the number of pills of ATX will be increased to 2 per day at the end of Week 1 of both Trials A and B. Subjects will remain on two capsules per day for the remaining 5 weeks of Trials A and B.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: atomoxetine — Subjects will receive ATX 40mg/d x 1 week, then 80mg/d x 5 weeks followed by a 4-week wash out period that is followed by an additional 6 weeks of treatment in the alternate condition. The 4-week washout period include a 4-day taper in the first week.
  Other Names: Strattera
  Arms: Atomoxetine
Drug: placebo — Subjects will receive placebo equivalent for 6 weeks followed by a 4-week wash out period that is followed by an additional 6 weeks of treatment in the alternate condition. The 4-week washout period include a 4-day taper in the first week.
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the efficacy of atomoxetine (ATX) treatment for the mild to moderate cognitive disturbances frequently experienced by women during the menopause transition. In addition, we seek to determine, using the Brown Attention Deficit Disorder Scale (BADDS), whether and to what degree peri- and early post-menopausal women experience cognitive disturbances which overlap with the impairments of executive function characteristic of adults with attention deficit disorder (ADHD).

DETAILED DESCRIPTION:
Decline in cognitive function, and in particular memory, is a frequent complaint for which menopausal women seek clinical intervention. While there is a wealth of preclinical evidence demonstrating the neuroprotective and cognitive enhancing role of estradiol (Wise et al., 1999; Jezierski & Sohrabji, 2001), recent publicity from the Women's Health Initiative Study has made gynecologists and menopausal women concerned about using estrogen therapy (ET) to address their cognitive complaints as well as other symptoms of menopause (WHI Writing Group, 2002). Decades of data suggesting that estrogen enhances cognitive function in women undergoing surgical or natural menopause (Sherwin et al., 1998) has been all but forgotten in the wake of the results of the WHI. Further, recent findings from a naturalistic study suggesting that having used estrogen replacement therapy for three years before the mean age of 70 years significantly reduced the risk of Alzheimer's Disease (AD; Zandi et al., 2002) did not receive sufficient attention in the lay press or in scientific circles to allay concerns. Most recently, conjugated equine estrogen plus medroxyprogesterone acetate (PremPro®) use daily is associated with a small increased risk for dementia (Schumaker et al., 2003).

Now that clinicians and women have become hesitant to utilize ET, they find themselves between the proverbial rock and a hard place as there have been no studies demonstrating efficacy of any other agent in the treatment of mild to moderate cognitive difficulties in healthy non-demented menopausal women. Thus, it is timely and crucial to investigate other pharmacologic strategies aimed at improving cognitive function in this population.

Interestingly, many of the cognitive complaints detected in menopausal women including, short-term memory, organization of tasks, sustaining focus and concentration, and regulating emotions, overlap with symptoms frequently reported by adults with ADHD (Warga, 1999; Brown, 2000). That ATX has demonstrated efficacy in the treatment of ADHD provides a compelling rationale for investigating the treatment of menopause-related declines in memory and cognitive function. Thus, this will be the first double-blind, placebo-controlled, cross-over clinical trial to obtain preliminary data for the efficacy of ATX in the treatment of mild to moderate cognitive disturbances in menopause aged women. Women who are in the early menopause have been chosen for this study as clinical and preclinical data suggest that long periods of hypoestrogenism may be associated with poorer response to intervention with ET. Therefore, we believe that this population may be more likely to respond to treatment with ATX than women who have been postmenopausal for many years.

ELIGIBILITY:
Inclusion Criteria:

* Menopausal subjects between the ages of 45 and 60 years;
* Physically healthy with no major medical illnesses;
* No history within the past 5 years of a DSM-IV psychiatric or substance abuse diagnosis by structured diagnostic interview (SCID);
* Subjects will be determined to be either peri or post-menopausal;
* Subjects must be within 5 years of their last menstrual period;
* Subjective report of cognitive disturbances of at least mild to moderate severity;
* All subjects must be of at least average intelligence as determined using the Wechsler Abbreviated Scale of Intelligence (WASI).

Exclusion Criteria:

* Clinical evidence of dementia and/or signs of dementia on the Mini-Mental Status Exam (MMSE score of <22);
* History of familial dementia;
* Use of any psychotropic medication within the previous 6 months;
* Use of any estrogen replacement therapy within the previous 6 months;
* Current pregnancy;
* Signs of an unstable medical or neurological disorder.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2004-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia N Epperson, MD, Principal Investigator — Yale University School of Medicine, Department of Psychiatry
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Background] Jezierski MK, Sohrabji F. Neurotrophin expression in the reproductively senescent forebrain is refractory to estrogen stimulation. Neurobiol Aging. 2001 Mar-Apr;22(2):309-19. doi: 10.1016/s0197-4580(00)00230-x. PMID 11182481
- [Background] Sherwin BB. Estrogen and cognitive functioning in women. Proc Soc Exp Biol Med. 1998 Jan;217(1):17-22. doi: 10.3181/00379727-217-44200. PMID 9421202
- [Background] Shumaker SA, Legault C, Rapp SR, Thal L, Wallace RB, Ockene JK, Hendrix SL, Jones BN 3rd, Assaf AR, Jackson RD, Kotchen JM, Wassertheil-Smoller S, Wactawski-Wende J; WHIMS Investigators. Estrogen plus progestin and the incidence of dementia and mild cognitive impairment in postmenopausal women: the Women's Health Initiative Memory Study: a randomized controlled trial. JAMA. 2003 May 28;289(20):2651-62. doi: 10.1001/jama.289.20.2651. PMID 12771112
- [Background] Wise PM, Smith MJ, Dubal DB, Wilson ME, Krajnak KM, Rosewell KL. Neuroendocrine influences and repercussions of the menopause. Endocr Rev. 1999 Jun;20(3):243-8. doi: 10.1210/edrv.20.3.0364. PMID 10368769
- [Background] Zandi PP, Carlson MC, Plassman BL, Welsh-Bohmer KA, Mayer LS, Steffens DC, Breitner JC; Cache County Memory Study Investigators. Hormone replacement therapy and incidence of Alzheimer disease in older women: the Cache County Study. JAMA. 2002 Nov 6;288(17):2123-9. doi: 10.1001/jama.288.17.2123. PMID 12413371

RESULTS

PARTICIPANT FLOW:
Groups:
- Atomoxetine Then Placebo; Placebo Then Atomoxetine: Subjects were enrolled into a double-blind, placebo-controlled cross over study where they will receive ATX 40mg/d x 1 week, then 80mg/d x 5 weeks or placebo (PBO) for 6 weeks, followed by a 4-week wash out period that is followed by an additional 6 weeks of treatment in the alternate condition. The 4-week washout period include a 4-day taper in the first week. Subjects will be instructed to take one capsule of ATX 40mg/d or placebo per day. If tolerated, the number of pills of ATX will be increased to 2 per day at the end of Week 1 of both Trials A and B. Subjects will remain on two capsules per day for the remaining 5 weeks of Trials A and B.
Period: First Intervention (6 Weeks)
Arm/Group | Atomoxetine Then Placebo | Placebo Then Atomoxetine
Started | 8 | 8
Completed | 8 | 6
Not Completed | 0 | 2
Not completed — Never started study | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Second Intervention (6 Weeks)
Arm/Group | Atomoxetine Then Placebo | Placebo Then Atomoxetine
Started | 8 | 6
Completed | 8 | 4
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Population: Participants who had at least one post randomization visit.
Groups:
- All Study Participants: Subjects were enrolled into a double-blind, placebo-controlled cross over study where they will receive ATX 40mg/d x 1 week, then 80mg/d x 5 weeks or placebo (PBO) for 6 weeks, followed by a 4-week wash out period that is followed by an additional 6 weeks of treatment in the alternate condition. The 4-week washout period include a 4-day taper in the first week. Subjects will be instructed to take one capsule of ATX 40mg/d or placebo per day. If tolerated, the number of pills of ATX will be increased to 2 per day at the end of Week 1 of both Trials A and B. Subjects will remain on two capsules per day for the remaining 5 weeks of Trials A and B.
Arm/Group | All Study Participants
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14
Years of education [Mean (Standard Deviation); unit: years] | 16.4 (3.2)
Months since last menstrual period [Mean (Standard Deviation); unit: months] | 29.3 (20.5)
Follicle stimulating hormone [Mean (Standard Deviation); unit: IU/L] | 76.0 (33.8)
Estradiol [Mean (Standard Deviation); unit: pg/mL] | 31.9 (32.9)
Brown attention deficit disorder scale [Mean (Standard Deviation); unit: units on a scale] — The total BADDS ranged from 0-120, with higher scores meaning greater problems with memory, attention and focus.
  units on a scale | 38.6 (20.2)
Participant characteristics [Count of Participants; unit: Participants] — OCP: Oral contraceptive pill; HT: Hormonal therapy
  Participants
    Perimenopausal | 4
    Postmenopausal | 10
    Previous OCP use | 11
    Previous HT use | 4

OUTCOME MEASURES:

1. Primary Outcome: Brown Attention Deficit Disorder Scale
Description: Raw scores for 5 clusters (organizing/activating, attention/concentration, alertness/effort/processing, managing affect interference, and working memory/recall) on the BADDS were converted to T scores which range from 50-99, with higher scores meaning greater impairment.
Time Frame: Baseline and after 6 weeks intervention
Population: Participants who completed both interventions.
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Baseline | Atomoxetine | Placebo
Number analyzed (Participants) | 12 | 12 | 12
T score
  organizing/activating | 60.7 (11.6) | 55.6 (8.9) | 56.3 (8.9)
  attention/concentration | 58.8 (8.7) | 52.1 (4.0) | 56.4 (7.1)
  alertness/effort/processing | 57.4 (10.0) | 54.2 (5.5) | 54.7 (7.9)
  managing affect interference | 55.3 (7.9) | 51.8 (4.5) | 51.6 (3.8)
  working memory/recall | 61.3 (10.0) | 52.4 (5.3) | 59.6 (10.3)

2. Primary Outcome: BADDS Total Score
Description: The total BADDS ranged from 0-120 with higher scores meaning greater problems with memory, attention and focus.
Time Frame: Baseline and after 6 weeks intervention
Population: Participants who had at least one post randomization visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline | Atomoxetine | Placebo
Number analyzed (Participants) | 14 | 14 | 14
units on a scale | 38.6 (20.2) | 25.5 (16.0) | 30.1 (16.0)

3. Secondary Outcome: Blood Pressure
Time Frame: Baseline and after 6 weeks intervention
Population: Participants who had least one post randomization visit.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Baseline | Atomoxetine | Placebo
Number analyzed (Participants) | 14 | 14 | 14
mm Hg
  systolic BP | 118.8 (12.5) | 116.7 (11.3) | 120.3 (8.5)
  diastolic BP | 74 (10.0) | 69.8 (7.7) | 70.7 (5.2)

4. Secondary Outcome: Heart Rate
Time Frame: Baseline and after 6 weeks intervention
Population: Participants who had at least one post randomization visit.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Baseline | Atomoxetine | Placebo
Number analyzed (Participants) | 14 | 14 | 14
beats/min | 63 (3.2) | 68.8 (8.2) | 66.3 (5.5)

5. Secondary Outcome: Weight
Time Frame: Baseline and after 6 weeks intervention
Population: Participants who had at least one post randomization visit.
Measure: Mean (Standard Deviation); unit: lb
Arm/Group | Baseline | Atomoxetine | Placebo
Number analyzed (Participants) | 14 | 14 | 14
lb | 160.1 (41.8) | 158.1 (44.4) | 159.8 (42.6)

ADVERSE EVENTS:
Time Frame: Up to 16 weeks study intervention
Arm/Group | Atomoxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 2/16 | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atomoxetine (N=16) | Placebo (N=16)
Nausea (Gastrointestinal disorders) | 2 | 1
increase in blood pressure (Cardiac disorders) | 1 | 0
racing heart (Cardiac disorders) | 0 | 1
dry mouth (General disorders) | 0 | 1
racing thoughts (Psychiatric disorders) | 0 | 1
insomnia (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No